CLINICAL TRIAL: NCT00315120
Title: A Randomized Controlled Trial of Osteopathic Manipulative Treatment and Ultrasound Physical Therapy for Chronic Low Back Pain
Brief Title: Osteopathic Health Outcomes in Chronic Low Back Pain (OSTEOPATHIC) Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of North Texas Health Science Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Osteopathic Heritage Foundations (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, John C. Licciardone, D.O., M.S., M.B.A., Director, Osteopathic Research Center, University of North Texas Health Science Center
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 06-02-20-1; K24AT002422 (NIH)
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Results first posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-05

CONDITIONS: Low Back Pain
Keywords: Randomized controlled trial; Low back pain; Spinal manipulative therapy; Spinal manipulation; Osteopathic manipulation; Osteopathic medicine; Physical therapy modalities
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Active OMT and active (UST) (Other): Subjects in this group received active osteopathic manipulation and active ultrasound physical therapy
  Interventions: Procedure: A. Active OMT and active UST
- B (Sham OMT and active UST) (Other): Subjects in this group received sham osteopathic manipulation and active ultrasound physical therapy
  Interventions: Procedure: B. Sham OMT and active UST
- C (Active OMT and sham UST) (Other): Subjects in this group received active osteopathic manipulation and sham ultrasound physical therapy
  Interventions: Procedure: C. Active OMT and sham UST
- D (Sham OMT and sham UST) (Other): Subjects in this group received sham osteopathic manipulation and sham ultrasound physical therapy
  Interventions: Procedure: D. Sham OMT and sham UST

INTERVENTIONS:
Procedure: A. Active OMT and active UST — Active osteopathic manipulation (OMT) and active ultrasound physical therapy (UST)
  Arms: A (Active OMT and active (UST)
Procedure: B. Sham OMT and active UST — Sham osteopathic manipulation (OMT) and active ultrasound physical therapy (UST)
  Arms: B (Sham OMT and active UST)
Procedure: C. Active OMT and sham UST — Active osteopathic manipulation (OMT) and sham ultrasound physical therapy (UST)
  Arms: C (Active OMT and sham UST)
Procedure: D. Sham OMT and sham UST — Sham osteopathic manipulation (OMT) and sham ultrasound physical therapy (UST)
  Arms: D (Sham OMT and sham UST)

SUMMARY:
The purpose of this study is to determine whether osteopathic manipulative treatment (a type of spinal manipulative therapy used by osteopathic physicians) and ultrasound physical therapy are effective in the treatment of chronic low back pain.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether osteopathic manipulative treatment (a type of spinal manipulative therapy used by osteopathic physicians) and ultrasound physical therapy are effective in the treatment of chronic low back pain. This study uses a 2X2 factorial design to test the hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Must give a positive response to the question: "Have you had low back pain constantly or on most days for the last three months?"
* Must identify the low back as the primary site of pain
* Must agree to not receive any of the following outside of the study during the period of participation: osteopathic manipulative treatment, chiropractic adjustment (including "mobilization" or "manipulation"), physical therapy
* Women must not be pregnant or plan to become pregnant during the period of study participation (a negative pregnancy test and willingness to maintain an acceptable method of contraception will be required)

Exclusion Criteria:

* History of any of the following conditions which may be underlying causes of low back symptoms: cancer, spinal osteomyelitis, spinal fracture, herniated disc, ankylosing spondylitis, cauda equina syndrome
* History of surgery involving the low back within the past year or planned low back surgery in the future
* History of receiving Workers' Compensation benefits within the past three months
* Involvement in current litigation relating to back problems
* Current pregnancy or plan to become pregnant during the course of participation in the study
* Any of the following that may limit a provider's choice of osteopathic manipulative treatment techniques or hamper compliance with the study protocol: angina or congestive heart failure symptoms that occur at rest or with minimal activity, history of a stroke or transient ischemic attack within the past year
* Any of the following that may represent potential contraindications to receiving ultrasound physical therapy: implantation of a cardiac pacemaker, implantation of artificial joints or other biomedical devices, active bleeding or infection in the low back, pregnancy
* Use of intravenous, intramuscular, or oral corticosteroids within the past month
* History of osteopathic manipulative treatment, chiropractic adjustment, or physical therapy within the past three months or on more than three occasions during the past year
* Practitioner or student of any of the following: osteopathic medicine (D.O.) allopathic medicine (M.D.), chiropractic (D.C.), physical therapy

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2006-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C. Licciardone, DO, MS, MBA, Principal Investigator — The Osteopathic Research Center, University of North Texas Health Science Center at Fort Worth
Locations (1):
- The Osteopathic Research Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Licciardone JC, Brimhall AK, King LN. Osteopathic manipulative treatment for low back pain: a systematic review and meta-analysis of randomized controlled trials. BMC Musculoskelet Disord. 2005 Aug 4;6:43. doi: 10.1186/1471-2474-6-43. PMID 16080794
- [Background] Licciardone JC, King HH, Hensel KL, Williams DG. OSTEOPAThic Health outcomes in chronic low back pain: The OSTEOPATHIC Trial. Osteopath Med Prim Care. 2008 Apr 25;2:5. doi: 10.1186/1750-4732-2-5. PMID 18439282
- [Background] Clinical Guideline Subcommittee on Low Back Pain; American Osteopathic Association. American Osteopathic Association guidelines for osteopathic manipulative treatment (OMT) for patients with low back pain. J Am Osteopath Assoc. 2010 Nov;110(11):653-66. PMID 21135197
- [Background] Licciardone JC, Gatchel R, Dagenais S. Assessment and management of back pain. JAMA Intern Med. 2014 Mar;174(3):478-9. doi: 10.1001/jamainternmed.2013.13692. No abstract available. PMID 24590092
- [Background] Licciardone JC. Osteopathic manual treatment and ultrasound therapy for chronic low back pain: an illustration of osteopathic semantic confusion. Author reply. J Am Osteopath Assoc. 2013 Sep;113(9):661-2. doi: 10.7556/jaoa.2013.031. No abstract available. PMID 24133757
- [Background] Licciardone JC. Systematic review and meta-analysis conclusions relating to osteopathic manipulative treatment for low back pain remain valid and well accepted. J Bodyw Mov Ther. 2013 Jan;17(1):2-4. doi: 10.1016/j.jbmt.2012.10.003. Epub 2012 Nov 16. No abstract available. PMID 23294676
- [Background] Licciardone JC. Osteopathic manipulative treatment in patients with low back pain. Clin Rheumatol. 2011 Jun;30(6):871-2; author reply 873. doi: 10.1007/s10067-011-1739-9. Epub 2011 Apr 15. No abstract available. PMID 21494808
- [Result] Licciardone JC, Kearns CM, Minotti DE. Outcomes of osteopathic manual treatment for chronic low back pain according to baseline pain severity: results from the OSTEOPATHIC Trial. Man Ther. 2013 Dec;18(6):533-40. doi: 10.1016/j.math.2013.05.006. Epub 2013 Jun 10. PMID 23759340
- [Result] Licciardone JC, Kearns CM, Hodge LM, Minotti DE. Osteopathic manual treatment in patients with diabetes mellitus and comorbid chronic low back pain: subgroup results from the OSTEOPATHIC Trial. J Am Osteopath Assoc. 2013 Jun;113(6):468-78. PMID 23739758
- [Result] Licciardone JC, Minotti DE, Gatchel RJ, Kearns CM, Singh KP. Osteopathic manual treatment and ultrasound therapy for chronic low back pain: a randomized controlled trial. Ann Fam Med. 2013 Mar-Apr;11(2):122-9. doi: 10.1370/afm.1468. PMID 23508598
- [Result] Licciardone JC, Gatchel RJ, Kearns CM, Minotti DE. Depression, somatization, and somatic dysfunction in patients with nonspecific chronic low back pain: results from the OSTEOPATHIC Trial. J Am Osteopath Assoc. 2012 Dec;112(12):783-91. PMID 23212429
- [Result] Licciardone JC, Kearns CM, Hodge LM, Bergamini MV. Associations of cytokine concentrations with key osteopathic lesions and clinical outcomes in patients with nonspecific chronic low back pain: results from the OSTEOPATHIC Trial. J Am Osteopath Assoc. 2012 Sep;112(9):596-605. doi: 10.7556/jaoa.2012.112.9.596. PMID 22984233
- [Result] Licciardone JC, Kearns CM. Somatic dysfunction and its association with chronic low back pain, back-specific functioning, and general health: results from the OSTEOPATHIC Trial. J Am Osteopath Assoc. 2012 Jul;112(7):420-8. PMID 22802542
- [Result] Licciardone JC. Short-term dosing of manual therapies for chronic low back pain. Spine J. 2014 Jun 1;14(6):1085-6. doi: 10.1016/j.spinee.2013.12.015. Epub 2013 Dec 20. No abstract available. PMID 24361999
- [Result] Licciardone JC, Kearns CM, Crow WT. Changes in biomechanical dysfunction and low back pain reduction with osteopathic manual treatment: results from the OSTEOPATHIC Trial. Man Ther. 2014 Aug;19(4):324-30. doi: 10.1016/j.math.2014.03.004. Epub 2014 Mar 18. PMID 24704126
- [Result] Licciardone JC. The OSTEOPATHIC trial demonstrates significant improvement in patients with chronic low back pain as manifested by decreased prescription rescue medication use. J Am Osteopath Assoc. 2014 Jul;114(7):528-9. doi: 10.7556/jaoa.2014.103. No abstract available. PMID 25002440
- [Result] Licciardone JC, Aryal S. Clinical response and relapse in patients with chronic low back pain following osteopathic manual treatment: results from the OSTEOPATHIC Trial. Man Ther. 2014 Dec;19(6):541-8. doi: 10.1016/j.math.2014.05.012. Epub 2014 Jun 5. PMID 24965494
- [Derived] Licciardone JC, Gatchel RJ, Aryal S. Targeting Patient Subgroups With Chronic Low Back Pain for Osteopathic Manipulative Treatment: Responder Analyses From a Randomized Controlled Trial. J Am Osteopath Assoc. 2016 Mar;116(3):156-68. doi: 10.7556/jaoa.2016.032. PMID 26927909
- [Derived] Licciardone JC, Gatchel RJ, Aryal S. Recovery From Chronic Low Back Pain After Osteopathic Manipulative Treatment: A Randomized Controlled Trial. J Am Osteopath Assoc. 2016 Mar;116(3):144-55. doi: 10.7556/jaoa.2016.031. PMID 26927908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 455 participants were recruited from the Dallas-Fort Worth, Texas metroplex from August 2006 to September 2010 through newspaper advertisements, community agencies, and medical clinics, excluding OMT specialty clinics.
Pre-assignment Details: Participants were randomized after their study eligibility was confirmed by both telephonic and clinical screening examinations.
Groups:
- OMT + UST: Active osteopathic manipulation and active ultrasound physical therapy
- Sham OMT + UST: Sham osteopathic manipulation and active ultrasound physical therapy
- OMT + Sham UST: Active osteopathic manipulation and sham ultrasound physical therapy
- Sham OMT + Sham UST: Sham osteopathic manipulation and sham ultrasound physical therapy
Period: Overall Study
Arm/Group | OMT + UST | Sham OMT + UST | OMT + Sham UST | Sham OMT + Sham UST
Started | 115 | 118 | 115 | 107
Completed | 115 | 118 | 115 | 107
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OMT + UST | Sham OMT + UST | OMT + Sham UST | Sham OMT + Sham UST | Total
Number analyzed (Participants) | 115 | 118 | 115 | 107 | 455
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 111 | 117 | 112 | 105 | 445
  >=65 years | 4 | 1 | 3 | 2 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.50 (13.05) | 39.19 (11.90) | 41.97 (12.58) | 41.38 (12.99) | 40.74 (12.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 68 | 78 | 72 | 284
  Male | 49 | 50 | 37 | 35 | 171
Region of Enrollment [Number; unit: participants]
  United States | 115 | 118 | 115 | 107 | 455

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analogue Scale Score for Pain Over 12 Weeks (OMT vs Sham OMT)
Description: Comparison of the number (proportion) of participants in each study group who achieve a substantial improvement in low back pain over 12 weeks as determined by at least a 40-mm reduction (-40 mm) on the visual analogue scale score for pain compared with the baseline score. Changes in the visual analogue scale scores for pain over 12 weeks may potentially range from a 100-mm reduction (-100 mm) to a 100-mm increase (+100). Any reduction (negative score) represents an improvement in low back pain (i.e., a "better" outcome), while any increase (positive score) represents a worsening of low back pain (i.e., a "worse" outcome). However, only those "better" outcomes represented by change scores less than or equal to -40 mm are considered to represent substantial improvement in low back pain, which is the primary outcome measure of this study. For analyses wherein floor effects are important, the 40-mm reduction threshold for substantial improvement may be replaced by 50% reduction (-50%).
Time Frame: 12 weeks
Measure: Number; unit: participants
Groups:
- Active OMT: Active osteopathic manipulation
- Sham OMT: Sham osteopathic manipulation
Arm/Group | Active OMT | Sham OMT
Number analyzed (Participants) | 230 | 225
participants | 40 | 20
Statistical Analysis 1: Comparison: Active OMT vs Sham OMT; Test type: Superiority or Other; p = 0.007, Chi-squared; Response ratio = 2.0, 95% CI 2-sided [1.2 to 3.2]

2. Secondary Outcome: Roland Morris Disability Questionnaire (OMT and Sham OMT - Week 4)
Description: Overall scores range from 0 to 24, which higher scores representing greater deficits in back-specific functioning.
Time Frame: 4 weeks
Population: Week 4 Data
Measure: Median (Inter-Quartile Range); unit: RMDQ Scale
Arm/Group | Active OMT | Sham OMT
Number analyzed (Participants) | 230 | 225
RMDQ Scale | 4 [2 to 8] | 5 [2 to 9]

3. Secondary Outcome: Roland Morris Disability Questionnaire (OMT and Sham OMT - Week 8)
Description: Overall scores range from 0 to 24, which higher scores representing greater deficits in back-specific functioning.
Time Frame: 8 weeks
Population: Week 8 Data
Measure: Median (Inter-Quartile Range); unit: RMDQ Scale
Arm/Group | Active OMT | Sham OMT
Number analyzed (Participants) | 230 | 225
RMDQ Scale | 3 [1 to 7] | 3 [2 to 8]

4. Secondary Outcome: Roland Morris Disability Questionnaire (OMT and Sham OMT - Week 12)
Description: Overall scores range from 0 to 24, which higher scores representing greater deficits in back-specific functioning.
Time Frame: 12 weeks
Population: Week 12 Data
Measure: Median (Inter-Quartile Range); unit: RMDQ Scale
Arm/Group | Active OMT | Sham OMT
Number analyzed (Participants) | 230 | 225
RMDQ Scale | 2 [1 to 6] | 3 [1 to 7]

5. Secondary Outcome: Roland Morris Disability Questionnaire (UST and Sham UST - Week 4)
Description: Overall scores range from 0 to 24, which higher scores representing greater deficits in back-specific functioning.
Time Frame: 4 weeks
Population: Week 4 Data
Measure: Median (Inter-Quartile Range); unit: RMDQ Scale
Groups:
- Active UST: Active ultrasound physical therapy
- Sham UST: Sham ultrasound physical therapy
Arm/Group | Active UST | Sham UST
Number analyzed (Participants) | 233 | 222
RMDQ Scale | 4 [2 to 9] | 5 [2 to 9]

6. Primary Outcome: Change in Visual Analogue Scale Score for Pain Over 12 Weeks (Active UST vs Sham UST)
Description: as for outcome 1
Time Frame: 12 weeks
Measure: Number; unit: participants
Groups:
- Active UST: Active ultrasound therapy
- Sham UST: Sham ultrasound therapy
Arm/Group | Active UST | Sham UST
Number analyzed (Participants) | 233 | 222
participants | 32 | 28
Statistical Analysis 1: Comparison: Active UST vs Sham UST; Test type: Superiority or Other; p = 0.72, Chi-squared; Response ratio = 1.1, 95% CI 2-sided [0.7 to 1.7]

7. Secondary Outcome: Roland Morris Disability Questionnaire (UST and Sham UST - Week 8)
Description: Overall scores range from 0 to 24, which higher scores representing greater deficits in back-specific functioning.
Time Frame: 8 weeks
Population: Week 8 Data
Measure: Median (Inter-Quartile Range); unit: RMDQ Scale
Arm/Group | Active UST | Sham UST
Number analyzed (Participants) | 233 | 222
RMDQ Scale | 3 [1 to 8] | 4 [1 to 7]

8. Secondary Outcome: Roland Morris Disability Questionnaire (UST and Sham UST - Week 12)
Description: Overall scores range from 0 to 24, which higher scores representing greater deficits in back-specific functioning.
Time Frame: 12 weeks
Population: Week 12 Data
Measure: Median (Inter-Quartile Range); unit: RMDQ Scale
Arm/Group | Active UST | Sham UST
Number analyzed (Participants) | 233 | 222
RMDQ Scale | 3 [1 to 7] | 3 [1 to 7]

9. Secondary Outcome: Medical Outcomes Study SF-36 Health Survey (OMT and Sham OMT - Week 4)
Description: The general health scale ranges from 0 to 100, with higher scores representing better general health.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: SF-36 General Health Score
Arm/Group | Active OMT | Sham OMT
Number analyzed (Participants) | 230 | 225
SF-36 General Health Score | 71 [55 to 82] | 72 [52 to 86]

10. Secondary Outcome: Medical Outcomes Study SF-36 Health Survey (OMT and Sham OMT - Week 8)
Description: The general health scale ranges from 0 to 100, with higher scores representing better general health.
Time Frame: 8 weeks
Measure: Median (Inter-Quartile Range); unit: SF-36 General Health Score
Arm/Group | Active OMT | Sham OMT
Number analyzed (Participants) | 230 | 225
SF-36 General Health Score | 72 [57 to 85] | 72 [52 to 85]

11. Secondary Outcome: Medical Outcomes Study SF-36 Health Survey (OMT and Sham OMT - Week 12)
Description: The general health scale ranges from 0 to 100, with higher scores representing better general health.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: SF-36 General Health Score
Arm/Group | Active OMT | Sham OMT
Number analyzed (Participants) | 230 | 225
SF-36 General Health Score | 72 [52 to 87] | 72 [57 to 87]

12. Secondary Outcome: Medical Outcomes Study SF-36 Health Survey (UST and Sham UST - Week 4)
Description: The general health scale ranges from 0 to 100, with higher scores representing better general health.
Time Frame: 4 Weeks
Measure: Median (Inter-Quartile Range); unit: SF-36 General Health Score
Arm/Group | Active UST | Sham UST
Number analyzed (Participants) | 233 | 222
SF-36 General Health Score | 72 [54 to 87] | 72 [52 to 82]

13. Secondary Outcome: Medical Outcomes Study SF-36 Health Survey (UST and Sham UST - Week 8)
Description: The general health scale ranges from 0 to 100, with higher scores representing better general health.
Time Frame: 8 Weeks
Measure: Median (Inter-Quartile Range); unit: SF-36 General Health Score
Arm/Group | Active UST | Sham UST
Number analyzed (Participants) | 233 | 222
SF-36 General Health Score | 72 [54 to 85] | 72 [57 to 85]

14. Secondary Outcome: Medical Outcomes Study SF-36 Health Survey (UST and Sham UST - Week 12)
Description: The general health scale ranges from 0 to 100, with higher scores representing better general health.
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: SF-36 General Health Score
Arm/Group | Active UST | Sham UST
Number analyzed (Participants) | 233 | 222
SF-36 General Health Score | 72 [52 to 87] | 74 [54 to 87]

15. Secondary Outcome: Work Disability (OMT and Sham OMT - Week 4)
Description: Number of participants who reported losing one or more work days in the past 4 weeks because of low back pain.
Time Frame: 4 weeks
Population: Lost 1 or more days of work in past 4 weeks because of low back pain.
Measure: Number (95% Confidence Interval); unit: Participants who reported lost work days
Arm/Group | Active OMT | Sham OMT
Number analyzed (Participants) | 107 | 100
Participants who reported lost work days | 11 [4 to 17] | 14 [7 to 21]

16. Secondary Outcome: Work Disability (OMT and Sham OMT - Week 8)
Description: Number of participants who reported losing one or more work days in the past 4 weeks because of low back pain.
Time Frame: 8 weeks
Population: Lost 1 or more days of work in past 4 weeks because of low back pain.
Measure: Number (95% Confidence Interval); unit: Participants who reported lost work days
Arm/Group | Active OMT | Sham OMT
Number analyzed (Participants) | 108 | 103
Participants who reported lost work days | 7 [2 to 12] | 20 [12 to 28]

17. Secondary Outcome: Work Disability (OMT and Sham OMT - Week 12)
Description: Number of participants who reported losing one or more work days in the past 4 weeks because of low back pain.
Time Frame: 12 weeks
Population: Lost 1 or more days of work in past 4 weeks because of low back pain.
Measure: Number (95% Confidence Interval); unit: Participants who reported lost work days
Arm/Group | Active OMT | Sham OMT
Number analyzed (Participants) | 108 | 103
Participants who reported lost work days | 12 [5 to 18] | 8 [3 to 13]

18. Secondary Outcome: Work Disability (UST and Sham UST - Week 4)
Description: Number of participants who reported losing one or more work days in the past 4 weeks because of low back pain.
Time Frame: 4 weeks
Population: Lost 1 or more days of work in past 4 weeks because of low back pain.
Measure: Number (95% Confidence Interval); unit: Participants who reported lost work days
Arm/Group | Active UST | Sham UST
Number analyzed (Participants) | 110 | 97
Participants who reported lost work days | 18 [10 to 25] | 7 [2 to 12]

19. Secondary Outcome: Work Disability (UST and Sham UST - Week 8)
Description: Number of participants who reported losing one or more work days in the past 4 weeks because of low back pain.
Time Frame: 8 weeks
Population: Lost 1 or more days of work in past 4 weeks because of low back pain.
Measure: Number (95% Confidence Interval); unit: Participants who reported lost work days
Arm/Group | Active UST | Sham UST
Number analyzed (Participants) | 112 | 99
Participants who reported lost work days | 19 [11 to 27] | 8 [3 to 14]

20. Secondary Outcome: Work Disability (UST and Sham UST - Week 12)
Description: Number of participants who reported losing one or more work days in the past 4 weeks because of low back pain.
Time Frame: 12 weeks
Population: Lost 1 or more days of work in past 4 weeks because of low back pain.
Measure: Number (95% Confidence Interval); unit: Participants who reported lost work days
Arm/Group | Active UST | Sham UST
Number analyzed (Participants) | 112 | 99
Participants who reported lost work days | 14 [7 to 21] | 6 [1 to 11]

21. Secondary Outcome: Satisfaction With Back Care (OMT and Sham OMT - Week 4)
Description: Subjects who reported being very satisfied with back care
Time Frame: 4 weeks
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Active OMT | Sham OMT
Number analyzed (Participants) | 208 | 208
participants | 109 [96 to 123] | 71 [58 to 85]

22. Secondary Outcome: Satisfaction With Back Care (OMT and Sham OMT - Week 8)
Description: Subjects who reported being very satisfied with back care
Time Frame: 8 weeks
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Active OMT | Sham OMT
Number analyzed (Participants) | 213 | 213
participants | 129 [115 to 143] | 84 [70 to 98]

23. Secondary Outcome: Satisfaction With Back Care (OMT and Sham OMT - Week 12)
Description: Subjects who reported being very satisfied with back care
Time Frame: 12 weeks
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Active OMT | Sham OMT
Number analyzed (Participants) | 216 | 213
participants | 143 [130 to 158] | 92 [77 to 107]

24. Secondary Outcome: Satisfaction With Back Care (UST and Sham UST - Week 4)
Description: Subjects who reported being very satisfied with back care
Time Frame: 4 weeks
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Active UST | Sham UST
Number analyzed (Participants) | 210 | 206
participants | 87 [74 to 101] | 93 [78 to 107]

25. Secondary Outcome: Satisfaction With Back Care (UST and Sham UST - Week 8)
Description: Subjects who reported being very satisfied with back care
Time Frame: 8 weeks
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Active UST | Sham UST
Number analyzed (Participants) | 217 | 209
participants | 107 [93 to 122] | 106 [92 to 121]

26. Secondary Outcome: Satisfaction With Back Care (UST and Sham UST - Week 12)
Description: Subjects who reported being very satisfied with back care
Time Frame: 12 weeks
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Active UST | Sham UST
Number analyzed (Participants) | 219 | 210
participants | 120 [105 to 134] | 115 [101 to 130]

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- OMT + UST: Active osteopathic manipulation and active ultrasound therapy
- Sham OMT + UST: Sham osteopathic manipulation and active ultrasound therapy
- OMT + Sham UST: Active osteopathic manipulation and sham ultrasound therapy
- Sham OMT + Sham UST: Sham osteopathic manipulation and sham ultrasound therapy
Arm/Group | OMT + UST | Sham OMT + UST | OMT + Sham UST | Sham OMT + Sham UST
Serious Adverse Events (participants affected / at risk) | 1/115 | 2/118 | 5/115 | 1/107
Other Adverse Events (participants affected / at risk) | 6/115 | 5/118 | 4/115 | 3/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | OMT + UST (N=115) | Sham OMT + UST (N=118) | OMT + Sham UST (N=115) | Sham OMT + Sham UST (N=107)
Any serious adverse event according to Food and Drug Administration definition (General disorders) | 1 (1) | 2/115 (2) | 5 (5) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OMT + UST (N=115) | Sham OMT + UST (N=118) | OMT + Sham UST (N=115) | Sham OMT + Sham UST (N=107)
Any other adverse event (General disorders) | 6 (6) | 5 (5) | 4 (4) | 3 (3)

LIMITATIONS AND CAVEATS:
Co-morbid conditions, work disability and low back pain co-treatments were self reported by participants, but were not verified through medical or employment records. Missing data were imputed for 13% of participants at the final encounter.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No